CLINICAL TRIAL: NCT00434044
Title: Multicenter, Double-Blind, Placebo-Controlled, Randomized Phase III Study of Etanercept in the Treatment of Subjects With Ankylosing Spondylitis
Brief Title: Study Evaluating Etanercept in the Treatment of Subjects With Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A3-322
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

INTERVENTIONS:
Drug: Enbrel (etanercept)

SUMMARY:
This study will represent the sponsor's first controlled study of etanercept in Chinese subjects with Ankylosing Spondytitis (AS). This trial is designed to assess the safety and efficacy of etanercept compared to placebo in the treatment of patients with AS.

DETAILED DESCRIPTION:
Multicenter, double-blind, randomized, parallel and placebo-controlled outpatient study. The study consists of 2 parts: part A is a 6-week double-blind treatment period and part B is a 6-week open-label treatment period. During part A of the study, subjects will be randomly assigned to 1 of 2 treatment regimens: 2 etanercept 25 mg or placebo once weekly, administered subcutaneously (SC). After the completion of part A, all subjects will receive 2 etanercept 25 mg once weekly. The use of placebo as a control in part A is necessary to allow a valid comparison and to provide a quantitative assessment of effect.

ELIGIBILITY:
Inclusion Criteria:

1. Must be of Chinese ancestry and living in China.
2. Diagnosis of AS, as defined by Modified New York Criteria for Ankylosing Spondylitis.
3. Active AS at time of enrollment, defined by average of visual analog scale (VAS) values for duration and intensity of morning stiffness 30 and two of the following: VAS for patient global assessment 30; average of VAS for nocturnal and total pain 30; BASFI greater than or equal to 30 (all scores on a scale of 0 to 100).

Exclusion Criteria:

1. Complete ankylosis (fusion) of spine.
2. Previous treatment with etanercept, antibody to Tumor Necrosis Factor a (TNFa), or other TNFa inhibitors or other biologic agents.
3. Use of disease modifying antirheumatic drugs (DMARDs) other than hydroxychloroquine, sulphasalazine, and methotrexate within 4 weeks of baseline. Subjects treated with hydroxychloroquine, sulphasalazine, and methotrexate may continue these drugs during this study but doses must be held stable for 4 weeks before baseline examination and for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2007-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Assessment in Ankylosing Spondylitis (ASAS) response criteria 20% at week six.

SECONDARY OUTCOMES:
ASAS 20% response at all visits except week two. ASAS 50%, 70%, 40%, 5/6 responses at all visits.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer